CLINICAL TRIAL: NCT01407029
Title: A Prospective, Multicenter, Non-randomized, Clinical Outcomes Study of the R3® Acetabular System in Patients With Degenerative Hip Disease
Brief Title: R3® Acetabular System in Patients With Degenerative Hip Disease
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R3H01
Record Dates: First submitted 2010-08-06; First posted 2011-08-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-randomized, consecutive series, multicenter clinical study that will include patients who will have total hip replacement with the R3 Acetabular System.

DETAILED DESCRIPTION:
The study design was selected to assess the safety and effectiveness profile of the R3 Acetabular System in patients with degenerative joint disease requiring primary total hip replacement. A non¬-randomized, consecutive series of up to 158 patients will be enrolled, and a maximum of 8 sites will participate in the study. Each site is allowed to enroll up to 22 patients. When 158 patients are enrolled from all sites, enrollment will be stopped, regardless of the number contributed from each site. The clinical data from this study will be compared with a historical control. The study will include follow up through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of legal age to consent and skeletally mature.
* Patient requires primary total hip arthroplasty due to non-inflammatory degenerative joint disease (e.g. osteoarthritis, traumatic arthritis, avascular necrosis, and dysplasia/DDH)
* Patient has met an acceptable preoperative medical clearance and is free from or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk.
* The patient will be available for follow-up throughout the duration of the study.

Exclusion Criteria:

* Patient has active infection or sepsis (treated or untreated)
* Patient has any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery.
* Patient is pregnant or plans to become pregnant during the course of the study Patient has inadequate bone stock to support the device (e.g. severe osteopenia, family history of severe osteoporosis or osteopenia)
* Patient has inflammatory joint disease (e.g. rheumatoid arthritis)
* Patient has known moderate to severe renal insufficiency.
* Patient has a known or suspected metal sensitivity.
* Patient is immunosuppressed or receiving high doses of corticosteroids.
* Patient has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, or drug, alcohol abuse.
* Patient has BMI >40.
* Patient is a prisoner

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This clinical study can fulfill its objectives only if appropriate subjects are enrolled. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a particular patient is suitable.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Effectiveness will be measured using the Harris Hip Score (HHS), The HOOS self assessment questionnaire, and radiographic assessment. Radiographic measures consist of radiolucencies, component position changes, and bony changes. | 3 months, 1-5 years
  The objective of this study is to establish the safety and effectiveness of the R3 Acetabular System in primary total hip replacement.

SECONDARY OUTCOMES:
Adverse Events | Post Operative - 5 years
  All perioperative and postoperative device-related and surgical adverse events will be recorded during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Richard McCalden, MD, Principal Investigator — London Health Science Centre-University Hospital London Ontario; Colin Burnell, MD, Principal Investigator — Concordia Hospital, Winnipeg, Canada; James Comadoll, MD, Principal Investigator — Ro Medical Orthopedics, Salisbury NC; Richard Steinfeld, MD, Principal Investigator — Orthopaedic Center of Vero Beach, Vero Beach, FL; Craig Della Valle, MD, Principal Investigator — Rush University Medical Center; John Masonis, MD, Principal Investigator — OrthoCarolina Research Institute; Ryan Nunley, MD, Principal Investigator — Washington University Orthopedics; Michael Dunbar, MD, Principal Investigator — Halifax Infirmary
Locations (8):
- United States (5):
  - Orthopedic Center of Vero Beach, Vero Beach, Florida
  - Midwest Orthopedics at Rush University Medical Center, Chicago, Illinois
  - Washington University Orthopedics, St Louis, Missouri
  - Ortho Carolina, Charlotte, North Carolina
  - Novant Health Pinnacle Orthopedics, Salisbury, North Carolina
- Canada (3):
  - Concordia Hip and Knee Institute, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Health Science Center, London, Ontario

IPD SHARING:
Plan to Share IPD: No